CLINICAL TRIAL: NCT04221490
Title: Edwards EVOQUE Tricuspid Valve Replacement: Investigation of Safety and Clinical Efficacy After Replacement of Tricuspid Valve With Transcatheter Device
Brief Title: 2019-06 TRISCEND Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Valve Regurgitation; Heart Valve Diseases; Cardiovascular Diseases
Keywords: Tricuspid Regurgitation; Transcatheter; Replacement; Functional; Degenerative; Regurgitation; Valve Replacement; Cardiovascular Disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the Edwards EVOQUE Tricuspid Valve Replacement System
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — Replacement of the tricuspid valve through a transcatheter approach
  Other Names: Edwards EVOQUE Tricuspid Valve Replacement System

SUMMARY:
Prospective, multi-center study to assess safety and performance of the Edwards EVOQUE Tricuspid Valve Replacement System

DETAILED DESCRIPTION:
The study is a multi-center, prospective single arm study designed to evaluate the safety and performance of the Edwards EVOQUE Tricuspid Valve Replacement System.

ELIGIBILITY:
Key Inclusion Criteria:

* Functional or degenerative TR moderate or greater
* Symptomatic despite medical therapy or prior HF hospitalization from TR
* The Local Site Heart Team determines that the patient is appropriate for transcatheter tricuspid valve replacement

Key Exclusion Criteria:

* Tricuspid valve anatomic contraindications
* Need for emergent or urgent surgery or any planned cardiac surgery within the next 12 months
* Hemodynamic instability
* Refractory heart failure requiring advanced intervention
* Currently participating in another investigational study in which the patient has not reached a primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2029-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susheel Kodali, MD, Principal Investigator — Columbia University
Locations (20):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital Boston, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Irving Medical Center / NYPH, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Heart Hopsital Plano, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (3):
  - St. Paul's Hospital Vancouver, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval (IUCPQ-ULaval), Québec
- France (2):
  - CHU Bordeaux, Hôpital Cardiologique Haut Lévêque, Pessac
  - Clinique Pasteur, Toulouse
- InselSpital University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodali S, Hahn RT, Makkar R, Makar M, Davidson CJ, Puthumana JJ, Zahr F, Chadderdon S, Fam N, Ong G, Yadav P, Thourani V, Vannan MA, O'Neill WW, Wang DD, Tchetche D, Dumonteil N, Bonfils L, Lepage L, Smith R, Grayburn PA, Sharma RP, Haeffele C, Babaliaros V, Gleason PT, Elmariah S, Inglessis-Azuaje I, Passeri J, Herrmann HC, Silvestry FE, Lim S, Fowler D, Webb JG, Moss R, Modine T, Lafitte S, Latib A, Ho E, Goldberg Y, Shah P, Nyman C, Rodes-Cabau J, Bedard E, Brugger N, Sannino A, Mack MJ, Leon MB, Windecker S; the TRISCEND study investigators. Transfemoral tricuspid valve replacement and one-year outcomes: the TRISCEND study. Eur Heart J. 2023 Dec 7;44(46):4862-4873. doi: 10.1093/eurheartj/ehad667. PMID 37930776
- [Background] Kodali S, Hahn RT, George I, Davidson CJ, Narang A, Zahr F, Chadderdon S, Smith R, Grayburn PA, O'Neill WW, Wang DD, Herrmann H, Silvestry F, Elmariah S, Inglessis I, Passeri J, Lim DS, Salerno M, Makar M, Mack MJ, Leon MB, Makkar R; TRISCEND Investigators. Transfemoral Tricuspid Valve Replacement in Patients With Tricuspid Regurgitation: TRISCEND Study 30-Day Results. JACC Cardiovasc Interv. 2022 Mar 14;15(5):471-480. doi: 10.1016/j.jcin.2022.01.016. PMID 35272771

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards EVOQUE Tricuspid Valve Replacement System: Treatment with the Edwards EVOQUE Tricuspid Transcatheter Valve Replacement System
Period: At 30 Days Follow-up
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Started | 228
Completed | 215
Not Completed | 13
Not completed — Death | 7
Not completed — Physician Decision | 1
Not completed — Missed Visit | 4
Not completed — Exited for Other Reasons | 1
Period: At 6 Months Follow-up
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Started | 219
Completed | 194
Not Completed | 25
Not completed — Death | 9
Not completed — Missed Visit | 8
Not completed — Exited for Other Reasons | 8
Period: At 1 Year Follow-up
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Started | 202
Completed | 183
Not Completed | 19
Not completed — Death | 7
Not completed — Withdrawal by Subject | 2
Not completed — Missed Visit | 9
Not completed — Exited for Other Reasons | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants who received any amount of study drug
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 228
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.5 (7.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 165
  Not Applicable | 30
  Other | 9
NYHA Class [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    Class I | 3
    Class II | 66
    Class III | 152
    Class IV | 7
Tricuspid Valve Disease Etiology [Count of Participants; unit: Participants] — Underlying cause of tricupsid regurgitation
  Participants
    Primary (Degenerative, Organic, Structural, or Pacer-related) | 27
    Secondary (Functional or Non-structural) | 159
    Mixed | 32
    Indeterminate | 10

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Events (MAEs)
Description: Composite of major adverse events (MAE) defined as cardiovascular mortality, myocardial infarction, stroke, renal complications requiring unplanned dialysis or renal replacement therapy, severe bleeding, unplanned or emergency tricuspid valve re-intervention, major access site and vascular complications, major access site and vascular complications, and device-related pulmonary embolism at 30 days.
Time Frame: 30 Days
Population: Analysis includes patients who had an MAE or who were followed for at least 30 days. Patients may experience more than one MAE.
Measure: Count of Participants; unit: Participants
Groups:
- Edwards EVOQUE Tricuspid Valve Replacement System: Treatment with the Edwards EVOQUE Tricuspid Valve Replacement System
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 226
Participants | 38

2. Primary Outcome: Device Success
Description: Study device is deployed as intended and the delivery system is successfully retrieved as intended at the time of the patient's exit from the cardiac catheterization laboratory.
Time Frame: Intraprocedural
Population: Per device analysis as participants may have more than one device attempted
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
Number analyzed (Device) | 223
Device | 218

3. Primary Outcome: Procedure Success
Description: Device success without clinically significant paravalvular leak (PVL) on a transthoracic echocardiogram (assessed by the echo core lab) at time of discharge.
Time Frame: Discharge (Up to 7 days post procedure)
Population: The outcome is reported where data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 220
Participants | 212

4. Primary Outcome: Clinical Success
Description: Procedural success without MAEs at 30 days.
Time Frame: 30 Days
Population: The outcome is reported where data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 221
Participants | 179

5. Primary Outcome: Tricuspid Regurgitation Reduction
Description: Percentage of patients with at least 1 grade reduction in tricuspid regurgitation (TR) as measured by using a 5-grade classification system (mild, moderate, severe, massive, torrential). TR grade is assessed by an independent echocardiography core laboratory.
Time Frame: Discharge (Up to 7 days post procedure)
Population: The outcome is reported where data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 220
Participants | 220

6. Secondary Outcome: Tricuspid Regurgitation (TR) Grade
Description: Tricuspid regurgitation (TR) is measured by transthoracic echocardiogram (TTE) at each visit using a 5-grade classification system (mild, moderate, severe, massive, torrential). TR grade is assessed by an independent echocardiography core laboratory.
Time Frame: Baseline, 30 Days, 6 Months
Population: The outcome is reported where data are available. Follow-up in the TRISCEND study is ongoing. Results beyond 6 months will be posted after completion of full follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
Participants
  Baseline: None/Trace | 0
  Baseline: Mild | 0
  Baseline: Moderate | 25
  Baseline: Severe | 85
  Baseline: Massive | 54
  Baseline: Torrential | 58
  30 Days: number analyzed (Participants) | 208
  30 Days: None/Trace | 158
  30 Days: Mild | 45
  30 Days: Moderate | 5
  30 Days: Severe | 0
  30 Days: Massive | 0
  30 Days: Torrential | 0
  6 Months: number analyzed (Participants) | 180
  6 Months: None/Trace | 119
  6 Months: Mild | 59
  6 Months: Moderate | 2
  6 Months: Severe | 0
  6 Months: Massive | 0
  6 Months: Torrential | 0

7. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: NYHA Functional Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: Baseline, 30 Days, 6 Months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
Participants
  Baseline: Class I | 3
  Baseline: Class II | 65
  Baseline: Class III | 147
  Baseline: Class IV | 7
  30 Days: number analyzed (Participants) | 207
  30 Days: Class I | 53
  30 Days: Class II | 120
  30 Days: Class III | 31
  30 Days: Class IV | 3
  6 Months: number analyzed (Participants) | 180
  6 Months: Class I | 68
  6 Months: Class II | 96
  6 Months: Class III | 14
  6 Months: Class IV | 2

8. Secondary Outcome: Change in Six Minute Walk Test (6WMT) Distance
Description: Mean distance in meters walked during Six Minute Walk Test (6MWT) at each follow-up visit compared to baseline. 6MWT is a submaximal exercise test that measures the distance that a patient can walk on a flat surface in a period of 6 minutes.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
meters
  30 Days: number analyzed (Participants) | 183
  30 Days | 41.3 (85.63)
  6 Months: number analyzed (Participants) | 169
  6 Months | 52.6 (96.57)

9. Secondary Outcome: Change in Quality of Life Score as Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Mean KCCQ score at each follow-up visit compared to baseline. The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores range from 0-100, in which higher scores reflect better health status.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
points
  30 Days: number analyzed (Participants) | 202
  30 Days | 20.6 (24.71)
  6 Months: number analyzed (Participants) | 182
  6 Months | 27.2 (22.20)

10. Secondary Outcome: Change in Quality of Life as Measured by 36-Item Short Form Health Survey (SF-36) Mental Score
Description: Mean change in SF-36 mental score at each follow-up visit compared to baseline compared to baseline. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
points
  30 Days: number analyzed (Participants) | 188
  30 Days | 4.2 (13.38)
  6 Months: number analyzed (Participants) | 160
  6 Months | 6.2 (11.50)

11. Secondary Outcome: Change in Quality of Life as Measured by 36-Item Short Form Health Survey (SF-36) Physical Score
Description: Mean change in SF-36 physical score at each follow-up visit compared to baseline. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
points
  30 Days: number analyzed (Participants) | 188
  30 Days | 5.1 (8.46)
  6 Months: number analyzed (Participants) | 160
  6 Months | 6.7 (9.35)

12. Secondary Outcome: Change in Body Weight
Description: Mean change in body weight in kilograms at each follow-up visit compared to baseline.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
kilograms
  30 Days: number analyzed (Participants) | 205
  30 Days | -2.2 (4.92)
  6 Months: number analyzed (Participants) | 186
  6 Months | -2.1 (5.90)

13. Secondary Outcome: Change in Left Ankle Circumference
Description: Mean change in left ankle circumference in centimeters at each follow-up visit compared to baseline.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
centimeters
  30 Days: number analyzed (Participants) | 199
  30 Days | -0.80 (2.836)
  6 Months: number analyzed (Participants) | 175
  6 Months | -0.60 (2.439)

14. Secondary Outcome: Change in Right Ankle Circumference
Description: Mean change in right ankle circumference in centimeters at each follow-up visit compared to baseline.
Time Frame: 30 Days, 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
centimeters
  30 Days: number analyzed (Participants) | 198
  30 Days | -0.67 (2.839)
  6 Months: number analyzed (Participants) | 174
  6 Months | -0.52 (2.685)

15. Secondary Outcome: Edema Assessment By Visit
Description: The edema grading scale measures how quickly the dimple goes back to normal (rebound) after a pitting test. The scale includes:
  Grade 1: Immediate rebound with 0 to 2 millimeter (mm) pit. Grade 2: Less than 15-second rebound with 3 to 4 mm pit. Grade 3: Rebound greater than 15 seconds but less than 60 seconds with 5 to 6 mm pit.
  Grade 4: Rebound between 2 to 3 minutes with an 8 mm pit.
Time Frame: Baseline, 30 Days, 6 Months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
Number analyzed (Participants) | 222
Participants
  Baseline: Absent | 73
  Baseline: Grade 1+ | 83
  Baseline: Grade 2+ | 47
  Baseline: Grade 3+ | 19
  Baseline: Grade 4+ | 0
  30 Days: number analyzed (Participants) | 202
  30 Days: Absent | 98
  30 Days: Grade 1+ | 74
  30 Days: Grade 2+ | 20
  30 Days: Grade 3+ | 8
  30 Days: Grade 4+ | 2
  6 Months: number analyzed (Participants) | 182
  6 Months: Absent | 99
  6 Months: Grade 1+ | 68
  6 Months: Grade 2+ | 10
  6 Months: Grade 3+ | 5
  6 Months: Grade 4+ | 0

ADVERSE EVENTS:
Time Frame: 1 year follow up
Arm/Group | Edwards EVOQUE Tricuspid Valve Replacement System
All-Cause Mortality (participants affected / at risk) | 23/228
Serious Adverse Events (participants affected / at risk) | 148/228
Other Adverse Events (participants affected / at risk) | 99/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards EVOQUE Tricuspid Valve Replacement System (N=228)
Air embolism (Vascular disorders) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 14 (14)
Bradycardia (Cardiac disorders) | 10 (10)
Bundle branch block right (Cardiac disorders) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Carcinoid syndrome (Endocrine disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 7 (7)
Cardiac failure (Cardiac disorders) | 19 (23)
Cardiogenic shock (Cardiac disorders) | 4 (4)
Haemorrhage (Vascular disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Haematoma (Vascular disorders) | 6 (6)
Haemolytic anaemia (Blood and lymphatic system disorders) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 12 (12)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5)
Gout (Metabolism and nutrition disorders) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Medical device site erosion (General disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 4 (5)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Prosthetic cardiac valve regurgitation (General disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 15 (16)
Device embolisation (General disorders) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 (20)
Glaucoma (Eye disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Prosthetic cardiac valve thrombosis (General disorders) | 3 (3)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 9 (9)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Distributive shock (Vascular disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (8)
Death (General disorders) | 2 (2)
Endocarditis (Infections and infestations) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 17 (17)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Device dislocation (Product Issues) | 6 (6)
Hypertension (Vascular disorders) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1)
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (5)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 5 (5)
Right ventricular failure (Cardiac disorders) | 6 (7)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 4 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Retroperitoneal haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Vessel puncture site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal mass (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Shock haemorrhagic (Vascular disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards EVOQUE Tricuspid Valve Replacement System (N=228)
Bundle branch block right (Cardiac disorders) | 20 (20)
Acute kidney injury (Renal and urinary disorders) | 21 (22)
Anaemia (Blood and lymphatic system disorders) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (19)
Atrial fibrillation (Cardiac disorders) | 15 (15)
Cardiac failure (Cardiac disorders) | 16 (18)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 18 (18)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 12 (13)
Troponin increased (Investigations) | 16 (16)
Hypotension (Vascular disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT04221490/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04221490/SAP_001.pdf